CLINICAL TRIAL: NCT02471105
Title: IOP and Tolerability Study of Preserved Bimatoprost 0.1% or Tafluprost Unit Dose Preservative Free 15microgram/ml, in Patients With OHT or Glaucoma Suitable for Prostaglandin Therapy
Brief Title: Investigation of IOP and Tolerability of Bimatoprost 0.01% and Tafluprost Unit Dose Preservative Free 15 Microgram/ml
Acronym: SPORTII
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: S57304
Record Dates: First submitted 2015-03-31; First posted 2015-06-15 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Ocular Hypertension; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — tafluprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumigan 0.01% + Saflutan 15 µg/ml (Experimental): Bimatoprost 0.01 % Eye drops solution Topical use Once in the evening 3 months
  Interventions: Drug: Preserved Bimatoprost 0.01%; Drug: Tafluprost Unit Dose Preservative Free 15microgram/ml
- Saflutan 15 µg/ml + Lumigan 0.01% (Experimental): Tafluprost Unit Dose Preservative Free 15microgram/ml Eye drops solution Topical use Once in the evening 3 months
  Interventions: Drug: Preserved Bimatoprost 0.01%; Drug: Tafluprost Unit Dose Preservative Free 15microgram/ml

INTERVENTIONS:
Drug: Preserved Bimatoprost 0.01% — Eye drops solution Topical use Once in the evening 3 months
  Other Names: BIMMD; Lumigan 0.01 %
Drug: Tafluprost Unit Dose Preservative Free 15microgram/ml — Eye drops solution Topical use Once in the evening 3 months
  Other Names: TUDPF; Saflutan

SUMMARY:
This cross-over study will investigate the efficacy and safety of BIMMD and TUDPF in a clinical setting.

DETAILED DESCRIPTION:
* A prospective, randomized, investigator-masked, crossover comparison;
* Ocular hypertension or glaucoma (XFG or POAG) patients and who consent to participate will be enrolled in this study
* Patients will be scheduled for a screening visit IOP assessment (IOP measurements at 08:30, 12:30 and 16:30 (±1 hour).
* Patients who are on therapy at the screening visit and who consent to participate will undergo a washout period for 4 weeks (depending on therapy) before the baseline visit;
* Patient can under the washout period be given brinzolamide (Azopt) if needed, Azopt should then be discontinued 5 days before baseline visit;
* After the screening visit (and after wash-outperiod for treated patients) patients will be scheduled to undergo a baseline visit IOP assessment (IOP measurements at 08:30, 12:30 and 16:30 (± 1 hour with a minimum of 3 hours between readings) and will then be randomized for Period 1 to receive either BIMMD drops once in the evening (20:30) or TUDPF drops once in the evening (20:30) for 3 month
* After 3 month, patients will be switched for Period 2, to the opposite treatment (e.g. switched to either BIMMD or TUDPF) to be dosed in the evening;
* After another 3 months they will undergo the final evaluation of IOP levels and of tolerability;
* Intermediate safety visits may be scheduled at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* A patient suffering from ocular hypertension, XFG or POAG and needs treatment in both eyes
* Patient is at least 18 years
* Patient is able and willing to participate in the study for the whole duration of the follow up and is willing to sign the consent form.

Exclusion Criteria:

* Unwilling to sign informed consent;
* Younger than 18 years old;
* Ocular condition that are of safety concern and that can interfere with the study results;
* Visual field defects with an MD value above -15dB on either eye on Humphrey (or the equivalent in Octopus) and/or threatening fixation
* Contact lens wearer;
* Closed/barely open anterior chamber angles or history of acute angle closure on either eye as assessed by gonioscopy;
* Ocular surgery (other than glaucoma surgery) or argon laser trabeculoplasty within the past three months on either eye;
* Glaucoma surgery within the past 6 months on either eye;
* Ocular inflammation/infection occurring within three months prior to pre-trial visit on either eye;
* Concomitant topical ocular medication that can interfere with study medication on either eye;
* Known hypersensitivity to any component of the trial drug solutions;
* Other abnormal condition or symptom preventing the patient from entering the trial, according to the Investigator's judgement;
* Refractive surgery patients at any time;
* Women who are pregnant, are of childbearing potential and are not using adequate contraception or are nursing;
* Inability to adhere to treatment/visit plan;
* Have participated in any other Interventional clinical trial (i.e., requiring informed consent) involving an investigational drug within one month prior to pre-trial visit.
* History of COPD, asthma or heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the difference in mean IOP values between the 2 groups | 6 months

SECONDARY OUTCOMES:
the difference in IOP values between the groups in change from baseline IOP | month 3 and month 6
the difference in mean IOP between the 2 groups | month 3
the difference in IOP between the 2 groups at each timepoints | month 3 and month 6

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, Phd, Principal Investigator — UZ Leuven
Locations (7):
- Hommer Ophthalmology Institute, Vienna, Austria
- UZ Leuven, Leuven, Vlaams Brabant, Belgium
- Italy (2):
  - San Paolo Hospital, Milan
  - Bietti Foundation, Rome
- Clinical Research Centre Momorial A. de Rotschild, Geneva, Switzerland
- United Kingdom (2):
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - Western Eye Hospital, London

REFERENCES:
- [Derived] Lemmens S, Rossetti L, Oddone F, Sunaric-Megevand G, Hommer A, Vandewalle E, Francesca Cordeiro M, McNaught A, Montesano G, Stalmans I. Comparison of preserved bimatoprost 0.01% with preservative-free tafluprost: A randomised, investigator-masked, 3-month crossover, multicentre trial, SPORT II. Eur J Ophthalmol. 2021 Apr 5:11206721211006573. doi: 10.1177/11206721211006573. Online ahead of print. PMID 33818170